CLINICAL TRIAL: NCT04876365
Title: Real-World Effectiveness of PEGylated, Recombinant Antihemophilic Factor (Adynovate) Prophylaxis in Patients With Hemophilia A in Canada: A Retrospective, Intra-patient Comparison With a Before-After Design
Brief Title: A Study in Children, Teenagers and Adults With Severe Hemophilia A Who Switched From Other Factor VIII Treatments to Adynovate
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-660-4004; MACS-2020-061601 (Other: Takeda)
Record Dates: First submitted 2021-05-05; First posted 2021-05-06 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All participants diagnosed with severe hemophilia A previous received prophylaxis regimen for Standard Half-life/Extended Half-life Factor VIII (SHL/EHL-FVIII) products will be compared to after the participants switched to regular prophylaxis with Adynovate with at least 6 months follow up.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — This is a Non-Interventional Study.

SUMMARY:
The main aims of the study are to assess the safety profile of Adynovate as well as how well people respond to the preventive treatment with Adynovate.

This study is about reviewing and collecting data of the participants before and after the switch to Adynovate that are already available. No new information will be collected during this study. The total time for data collection in the study will be approximately 72 months (36 months before and 36 months after switching to Adynovate). Participants will not receive Adynovate as part of this study.

As participants are not treated in this study, they do not need to visit their doctor in addition to their normal visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants with severe hemophilia A.
* All age groups (less than [<] 12 and greater than [>] 12 years of age).
* Participant with greater than equal to (>=) 150 documented exposure days (EDs).
* Treated with Adynovate:

  * Having a PK analysis done/data available for post-hoc modeling
  * Having recorded clinical outcomes analysis: for > 6 months
* Treated with a SHL/EHL-FVIII product for at least six months before switching to Adynovate
* To qualify for the secondary objective participants will need to have a WAPPS study performed on Adynovate and on the SHL/EHL-FVIII they were treated before switching.

Exclusion Criteria:

* Any participant who meets any of the following criteria will not qualify for entry into the study:
* Participants with only on-demand Factor VIII (FVIII) use.
* Current presence of FVIII inhibitory antibodies. (Participants with a history of inhibitors, if any, will be considered for a sensitivity analysis).
* Diagnosis of other inherited or acquired hemostatic defect other than hemophilia A.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will comprise of participants of all ages receiving regular prophylactic treatment with Adynovate at a Canadian Hemophilia Treatment Center and registered in CBDR (Canadian Bleeding Registry).
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Time Spent With Factor Levels Above 0.01 IU/ml | approximately 72 months
  Percentage of time spent with factor levels above 0.01 (International units per milliliter [IU/ml], is calculated as: time spent with factor levels above 0.01 IU/ml/ total time in the study. The calculation will be performed by simulating, based on the infusions recorded in the treatment diaries and the individual PK profiles, all the times intervals between each infusion and the time at which the concentration of 0.01 IU/mL is reached, and the time between reaching the 0.01 IU/mL and the subsequent infusion.
Number of Participants With Adverse Events (AEs) | approximately 72 months
  An AEs is any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. Number of participants with AEs related to inhibitor development, thrombosis, death, infection, cancer and other will be reported.

SECONDARY OUTCOMES:
Percentage of Time Spent With Factor Levels Above 0.03 IU/ml | approximately 72 months
  Percentage of time spent with factor levels above 0.03 IU/ml, is calculated as: time spent with factor levels above 0.03 IU/ml/ total time in the study. The calculation will be performed by simulating, based on the infusions recorded in the treatment diaries and the individual.
Percentage of Time Spent With Factor Levels Above 0.05 IU/ml | approximately 72 months
  Percentage of time spent with factor levels above 0.05 IU/ml, is calculated as: time spent with factor levels above 0.05 IU/ml/ total time in the study. The calculation will be performed by simulating, based on the infusions recorded in the treatment diaries and the individual.
Terminal Half-life of Adynovate | approximately 72 months
  Terminal half-life will be estimated based on the individual Web-Accessible Population Pharmacokinetic Hemophilia Service (WAPPS) PK profile.
Clearance (Cl) of Adynovate | approximately 72 months
  Cl will be estimated based on the individual WAPPS PK profile.
Maximum Observed Drug Concentration (Cmax) of Adynovate | approximately 72 months
  Cmax is as estimated based on the individual WAPPS PK profile.
Area Under the Curve (AUC) of Adynovate | approximately 72 months
  AUC will be estimated based on the individual WAPPS PK profile.
Annualized Total Factor Consumption | approximately 72 months
  The total factor consumption will be measured on the infusion log, annualized and adjusted per body weight. Annualized FVIII concentrate consumption, adjusted per body weight, will be calculated as: total amount infused IU/ Weight (kilograms)*12/months of observation.
Annualized Total Factor Consumption for Bleeds | approximately 72 months
  The total factor consumption for bleeds will be measured on the infusion log, annualized and adjusted per body weight. Annualized FVIII concentrate consumption, adjusted per body weight, will be calculated as: total amount infused IU for bleeds/ Weight (kilograms)*12/months of observation.
Estimated Factor Consumption | approximately 72 months
  Estimated factor consumption, based on the prescribed treatment regimen, annualized and adjusted per body weight, is calculated as: total amount prescribed (IU)/week / Weight (kilograms)*52/weeks of observation.
Theoretical Factor Consumption | approximately 72 months
  Theoretical factor consumption, estimated based on the amount required to obtain specified factor level troughs (0.03 IU/mL, 0.10 IU/mL), annualized and adjusted per body weight, will be calculated as: estimated amount prescribed IU/week / Weight (kilograms)*52/weeks of observation.
Annualized Bleeding Rate (ABR) | approximately 72 months
  ABR will be calculated as: number of bleeds*12/months of observation.
Annualized Spontaneous Bleeding Rate (AsBR), | approximately 72 months
  AsBR will be calculated as: number of spontaneous bleeds*12/months of observation. A bleed is defined as spontaneous if it is not related to injury/trauma.
Annualized Joint Bleeding Rate (AjBR) | approximately 72 months
  AjBR will be calculated as: number of joint bleeds*12/months of observation. An acute joint bleed include some or all of the following: 'aura', pain, swelling, warmth of the skin over the joint, decreased range of motion and difficulty in using the limb compared with baseline or loss of function.
Hemophilia Joint Health Score (HJHS)- Total Score | approximately 72 months
  HJHS will be assessed based on the following components of the elbow, knee, and ankle joints: swelling, duration of swelling, muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain, and strength, together with an assessment of the global gait. The HJHS is a validated 11-item scoring tool based on radiologic and clinical evaluation, sensitive to detect early signs and minor changes. HJHS ranges from 0 to 124. Higher values in the HJHS represent worse situation for the participant.
Health-Related Quality of Life (HRQoL) Assessed by Patient-reported Outcome Burdens and Experiences (PROBE) Questionnaire | approximately 72 months
  The PROBE questionnaire is a tool for the assessment of patient-reported outcome, burdens and experiences. Until now, it has been used in persons living with hemophilia (PWH) and healthy controls. PROBE questionnaire consists of four major sections: demographic data, general health problems, hemophilia-related health problems and health-related quality of life. Scores range from 0-1, with a higher value indicating better health status.
HRQoL Assessed by EuroQoL Group 5-Dimension 5-Level Self-Report (EQ-5D-5L) | approximately 72 months
  The EQ-5D-5L descriptive system assesses health in five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). This part of the EQ-5D questionnaire provides a descriptive profile that can be used to generate a health state profile. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the participant rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Hamilton-Niagara Regional Hemophilia Treatment Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60990901ef0b71001e743c61